CLINICAL TRIAL: NCT06824818
Title: A Feasibility Trial of LHRH Agonist Discontinuation in Elderly Prostate Cancer Patients
Brief Title: Study to Assess the Feasibility of Stopping Prostate Cancer Treatment Early in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-1729
Record Dates: First submitted 2025-01-31; First posted 2025-02-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Elderly; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study follows a **single-group assignment** model, where all participants discontinue LHRH agonist therapy and are monitored for testosterone and PSA levels over 3 years to assess the feasibility of this approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- discontinuation of LHRH agonist therapy in elderly prostate cancer patients (Experimental)
  Interventions: Behavioral: LHRH Agonist Therapy Discontinuation

INTERVENTIONS:
Behavioral: LHRH Agonist Therapy Discontinuation — The intervention involves **discontinuing LHRH agonist therapy** in elderly prostate cancer patients who have been on long-term androgen deprivation therapy. Participants will be monitored for testosterone recovery and PSA levels over a period of up to 3 years.

SUMMARY:
This study seeks to identify if it is feasible to stop Luteinizing Hormone-Releasing Hormone (LHRH) Agonist Therapy in elderly men with prostate cancer. We hypothesize that elderly prostate cancer patients on long term androgen ablation with LHRH agonists will be permanently castrated and do not require ongoing LHRH agonist therapy. Participants will be monitored by testosterone testing throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer with >3 years of LHRH agonist therapy.
* Age ≥70 years.
* ECOG performance status ≤2
* Baseline testosterone of < 20 ng/ml
* No prior chemotherapy or Lu-PSMA (unless survival predictions are favorable).
* Ability to understand and sign informed consent.

Exclusion Criteria:

* none

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 155 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
feasibility of stopping LHRH agonist therapy | 12 months after discontinuing LHRH agonist therapy
  Fraction of patients maintaining castrate testosterone levels

SECONDARY OUTCOMES:
Patient interest in stopping treatment | End of enrollment (approximately 3 years after study start)
  Percentage of patients that decline participation in the study
Medication Impact | End of study (approximately 3 years after last participant is enrolled)
  Percentage of participants that start other prostate cancer treatments before starting or during the study
Impact on Testosterone Levels (12 months) | 12 months after last participant starts study
  Percentage of participants with testosterone levels <20 ng/ml
Impact on Testosterone Levels (36 months) | 36 months after last participant starts study
  Percentage of participants with testosterone levels <20 ng/ml
Health Care Savings | End of study (approximately 3 years after last participant is enrolled)
  Cost savings per participant measured by cost of the drug (e.g. how much was saved by participants not taking drug during the study period)
Visit Compliance | End of study (approximately 3 years after last participant is enrolled)
  Percentage of missed visits during study compared to number of routine visits missed in 12 month period prior to starting study

CONTACTS AND LOCATIONS:
Overall Officials: Nabiel Mir, MD, Study Chair — University of Chicago
Locations (2):
- United States (2):
  - The University of Illinois at Chicago (UIC), Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided